CLINICAL TRIAL: NCT01709942
Title: Use of Long Acting GnRH Antagonist to Prevent Ovarian HyperStimulation Syndrome (OHSS) in PCOS Women Undergoing COH for IVF
Brief Title: Use of Degarelix in Controlled Ovarian Hyperstimulation (COH) Protocol for Women With PoliCystic Ovarian Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre for Endocrinology and Reproductive Medicine, Italy (Network)
Responsible Party: Principal Investigator, Fabio Scarpellini, Principal Investigator, Centre for Endocrinology and Reproductive Medicine, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: C05
Record Dates: First submitted 2012-10-17; First posted 2012-10-18 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-04

CONDITIONS: PCOS; OHSS; INFERTILITY
Keywords: GnRH antagonist; PCOS; OHSS; COH; IVF
MeSH Terms: conditions — Infertility | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; cetrorelix

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- degarelix group (Experimental): group of patients treated with long acting GnRH antagonist
  Interventions: Drug: degarelix (long acting GnRH antagonist)
- Cetrorelix 0.25mg (Active Comparator): patients treated with gonadotropin and Cetrorelix ina flexible GnRH antagonist protocol
  Interventions: Drug: cetrorelix 0.25mg

INTERVENTIONS:
Drug: degarelix (long acting GnRH antagonist) — 20 mg of degarelix the first day of menstrual cycle before starting with gonadotrophins administration
  Other Names: Firmagon
  Arms: degarelix group
Drug: cetrorelix 0.25mg — 0.25mg of cetrorelix during treatment with gonadotrophins when estradiol levels were >300pg/ml
  Other Names: cetrotide
  Arms: Cetrorelix 0.25mg

SUMMARY:
In this study the effectiveness of degarelix, a long acting GnRH antagonist administered in a unique administration of 20 mg the first day of menstrual cycle, to prevent ovarian hyperstimulation syndrome (OHSS) in PCOS women at risk to develop OHSS.

DETAILED DESCRIPTION:
Women with PCOS are at risk to develop OHSS when stimulated with gonadotrophins for IVF. For this reason in this study the degarelix was tested in order to minimize the risk of OHSS as well as to improve the pregnancy rate in these patients. The use of long acting GnRH antagonist promotes a deep suppression of LH and consequently the activity of theca cells, which secrete androgens (the precursors of estradiol), and consequently the levels of estradiol remains low. Comparing the long acting GnRH antagonist at the first day of cycle with a flexible GnRH antagonist protocol in a group of patients with PCOS will be useful in order to establish the best way to perform controlled hyperstimulation in IVF cycles and minimize the risk of OHSS.

ELIGIBILITY:
Inclusion Criteria:

* women with PCOS
* previous OHSS
* Infertility

Exclusion Criteria:

* more than 38 years old
* Body mass index pore than 30
* other systemic diseases

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2012-11; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
PREGNANCY RATE | 6 MONTHS
  number of ongoing pregnancy obtained in the group
ovarian hyperstimulation syndrome rate | 6 MONTHS
  incidence of ovarian hyperstimulation syndrome in the groups

SECONDARY OUTCOMES:
implantation rate | 6 months
  number of implanted embryos divided for the number of transferred embryos

OTHER OUTCOMES:
number of mature oocytes | 6 months
  number of mature oocytes obtained in each patient

CONTACTS AND LOCATIONS:
Overall Officials: Marco Sbracia, MD, Study Chair — Centre for Endocrinology and Reproductive Medicine, Italy
Locations (1):
- Cerm-Hungaria, Rome, Italy

REFERENCES:
- [Result] Garcia-Velasco JA, Kupesic S, Pellicer A, Bourgain C, Simon C, Mrazek M, Devroey P, Arce JC. Follicular and endocrine profiles associated with different GnRH-antagonist regimens: a randomized controlled trial. Reprod Biomed Online. 2012 Feb;24(2):153-62. doi: 10.1016/j.rbmo.2011.10.016. Epub 2011 Nov 4. PMID 22197127